CLINICAL TRIAL: NCT01230177
Title: Enbrel Qw Special Investigation (Regulatory Post Marketing Commitment Plan)
Brief Title: Etanercept (Enbrel) Special Investigation (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801134
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Arthritis; Rheumatoid
MeSH Terms: conditions — Arthritis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Etanercept (genetical recombination): Among the patients with rheumatoid arthritis (only for patients with an inadequate response to prior conventional therapy), the patients who will have changed regimen from 10 mg twice a week administration to 25 mg once a week administration.
  Interventions: Drug: etanercept (genetical recombination)

INTERVENTIONS:
Drug: etanercept (genetical recombination) — 10 to 25 mg of etanercept (genetical recombination) reconstituted in 1 mL of water for injection (JP) administered twice weekly as a subcutaneous injection or 25 to 50 mg of etanercept (genetical recombination) administered once weekly as a subcutaneous injection, are usually the recommended dose for adults.
  Other Names: Enbrel

SUMMARY:
This survey is conducted to investigate safety and efficacy under the post marketed drug utilization on the patient with rheumatoid arthritis (only for patients with an inadequate response to prior conventional therapy) at the time of switching regimen from 10 mg twice a week administration to 25 mg once a week administration.

DETAILED DESCRIPTION:
Implemented as a Special Investigation by Central Registration System

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered etanercept in order to be enrolled in the survey
* Patients who have changed regimen from 10 mg twice a week administration to 25 mg once a week administration.

Exclusion Criteria:

* Patients who have been administered etanercept 50mg once a week
* Patients who have been administered etanercept 25mg once a week

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Among the patients with rheumatoid arthritis (only for patients with an inadequate response to prior conventional therapy), the patients who will have changed regimen from 10 mg twice a week administration to 25 mg once a week administration.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Taihaku Sakura Hospital, Sendai, Miyagi, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801134&StudyName=Etanercept%20%28Enbrel%29%20Special%20investigation%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept（Genetial Recombination）: Participants in whom the regimen of etanercept was changed from 10 mg twice weekly to 25 mg once weekly for the treatment of rheumatoid arthritis.
Period: Overall Study
Arm/Group | Etanercept（Genetial Recombination）
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Etanercept (Renetical Recombination): Participants in whom the regimen of etanercept was changed from 10 mg twice weekly to 25 mg once weekly for the treatment of rheumatoid arthritis.
Arm/Group | Etanercept (Renetical Recombination)
Number analyzed (Participants) | 3
Age, Customized [Number; unit: participants]
  <65 years | 0
  >=65 years | 3
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events
Description: Adverse events are defined as any unfavorable events, including clinically significant abnormal changes in laboratory test values, which develop in participants after the administration of etanercept regardless of the causal relationship to etanercept. The causal relationship between an adverse event and etanercept was evaluated by the sponsor.
Time Frame: 12 weeks
Population: The safety analysis population consisted of the participants in whom the regimen of etanercept was changed from 10 mg twice weekly to 25 mg once weekly for the treatment of rheumatoid arthritis.
Measure: Number; unit: participants
Arm/Group | Etanercept（Genetial Recombination）
Number analyzed (Participants) | 3
participants | 2

2. Primary Outcome: Disease Activity Score of 28 Joints (DAS28: 4/Erythrocyte Sedimentation Rate [ESR])
Description: DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hour) and PtGA of disease activity (participant rated arthritis activity assessment). Total score range: 0-9.4, higher score=more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (ESR) <2.6 = remission.
  DAS28-3 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hour). Total score range: 0-9.4, higher score=more disease activity. DAS28-3 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (ESR) <2.6 = remission.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Etanercept（Genetial Recombination）
Number analyzed (Participants) | 1
Score
  At 0 week | 3.55 (0)
  At 8 weeks | 2.72 (0)

3. Secondary Outcome: Physician's Assessment of Clinical Effect of Etanercept on the Symptoms of Rheumatoid Arthritis and Change in Laboratory Values
Description: On the basis of how well the clinical symptoms of rheumatoid arthritis were controlled at baseline, the physician assessed the clinical effect of etanercept in two grades: "effective" or "ineffective". To assess the clinical efficacy of etanercept, the degrees of the symptoms of rheumatoid arthritis and laboratory test values were compared between at baseline and at the 12th week of the investigation.
Time Frame: 12 weeks
Population: The efficacy analysis population consisted of the participants in whom the change in DAS28 (4/ESR and 3/ESR) was calculated. No descriptive statistic on the change in DAS28 (4/ESR and 3/ESR) was calculated due to a very small number of participants (n = 3).
Measure: Number; unit: participants
Arm/Group | Etanercept（Genetial Recombination）
Number analyzed (Participants) | 3
participants
  Effective | 3
  Ineffective | 0

4. Secondary Outcome: Physician's Assessment of Clinical Effect of Etanercept on the Symptoms of Rheumatoid Arthritis and Change in Laboratory Values
Description: as for outcome 3
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Etanercept（Genetial Recombination）
Number analyzed (Participants) | 3
participants
  Effective | 3
  Ineffective | 0

5. Primary Outcome: Change in Disease Activity Score of 28 Joints (DAS28: 4/Erythrocyte Sedimentation Rate [ESR])
Description: as for outcome 2
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept（Genetial Recombination）
Number analyzed (Participants) | 1
percent change
  At 0 week | 0 (0)
  At 8 weeks | -23.58 (0)

ADVERSE EVENTS:
Description: The frequency of treatment related adverse events during the study
Arm/Group | Etanercept（Genetial Recombination）
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept（Genetial Recombination） (N=3)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept（Genetial Recombination） (N=3)
Nasopharyngitis (Infections and infestations) | 2 (2)
Keratitis (Eye disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.